CLINICAL TRIAL: NCT01328574
Title: A Phase II Study of TRC105 in Adults With Advanced/Metastatic Urothelial Carcinoma
Brief Title: TRC105 in Adults With Advanced/Metastatic Urothelial Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Andrea Apolo, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110130; 11-C-0130
Record Dates: First submitted 2011-04-01; First posted 2011-04-04 (Estimated); Results first posted 2015-03-02 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Urothelial Carcinoma; Ureteral Neoplasms; Ureter Cancer; Neoplasm, Ureteral; Cancer of the Ureter
Keywords: Progression-Free Survival; Carcinoma of the Bladder; Cancer of the Renal Pelvis; Ureter Cancer; Survival; Bladder Cancer; Renal Pelvis Cancer; Urothelial Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Ureteral Neoplasms; Urinary Bladder Neoplasms | interventions — carotuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm - TRC105 in Urothelial Carcinoma (Experimental): TRC105 15 mg/kg/dose every two weeks
  Interventions: Drug: TRC105

INTERVENTIONS:
Drug: TRC105 — 15 mg/kg intravenously

SUMMARY:
Background:

- Urothelial cancer (tumors of the bladder, urethra, ureter, or renal pelvis) often responds initially to standard chemotherapy treatments, but frequently recurs and can often spread to other parts of the body. TRC105, an experimental drug that blocks the development of the new blood vessels needed for tumor growth, may be able to shrink or stabilize urothelial cancer tumors. TRC105 has been given previously to individuals with other types of cancer, and researchers are interested in determining its safety and effectiveness in treating urothelial cancer.

Objectives:

- To determine the safety and effectiveness of TRC105 as a treatment for metastatic urothelial cancer that has not responded to standard treatments.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with urothelial cancer that has spread to other parts of the body and has not responded to standard chemotherapy.

Design:

* Participants will be screened with a physical examination, medical history, blood tests, and tumor imaging studies.
* Participants will receive TRC105 intravenously once every 2 weeks on days 1 and 15 of a 28-day treatment cycle. The first dose of TRC105 will be given over a 4-hour period; participants who do not have side effects may receive the next dose over 2 hours. If the second dose is tolerated, subsequent doses can be given over at least 1 hour.
* To help prevent known side effects of TRC105, participants will take two doses (one in the morning and one in the evening) of the steroid dexamethasone on the day before each infusion is scheduled. Participants may have additional dexamethasone 30 minutes before infusion, and may have the infusion slowed or stopped to adjust for side effects.
* Participants will be monitored with blood samples, physical examinations, and tumor imaging studies through the cycles of treatment.
* Participants will continue to take TRC105 for as long as the treatment is effective against the cancer and as long as the side effects are not severe enough to stop treatment.

DETAILED DESCRIPTION:
BACKGROUND:

* In the United States, urothelial carcinoma (UC) of the bladder is the 4th most common malignancy in men and the 9th most common in women with an estimated 70,980 new cases and 14,330 deaths in the year 2009. Although it is chemosensitive with response proportions of over 50% with conventional cytotoxic regimens, the response durations are short and the median survival of patients with metastatic disease is approximately 14 months.
* TRC105 is a genetically engineered human/murine chimeric monoclonal antibody that inhibits angiogenesis and tumor growth via endothelial cell growth inhibition and apoptosis. TRC105 is directed against human CD105 (endoglin), an angiogenic membrane protein that is highly expressed on proliferating vasculature in solid tumors and up-regulated following anti-VEGF (vascular endothelial growth factor) therapy. Clinical studies in bladder cancer with anti-angiogenic agents have shown anti-tumor activity.
* TRC105 targets a unique mechanism for tumor angiogenesis, through modification of CD105 signaling. In patients with advanced bladder cancer that have progressed through standard chemotherapy and have no further life prolonging therapeutic options, use of this novel angiogenesis inhibitor may improve outcomes.

OBJECTIVES:

* To measure PFS (progression free survival) of TRC105 as determined by RECIST (Response Evaluation Criteria in Solid Tumors) v1.1
* To determine the safety and toxicity of TRC105 in this patient population.
* In addition, in a preliminary fashion, response rate and overall survival of patients with metastatic urothelial carcinoma of the bladder treated with TRC105 will be estimated.

ELIGIBILITY:

* Adults with progressive advanced/metastatic urothelial carcinoma that have progressed despite treatment with prior cytotoxic chemotherapy.
* Subjects must have received at least one prior cytotoxic agent (which must have included at least one of the following: cisplatin, carboplatin, paclitaxel, docetaxel, or gemcitabine).

DESIGN:

* TRC105 will be administered at a dose of 15 mg/kg intravenously every two weeks, on days 1 and 15 of each 28 day cycle.
* Patients may continue on study as long as they are tolerating therapy and are free of disease progression.
* The study will be conducted as a two-stage optimal design (Simon 1989). With alpha=0.10 and beta=0.10 as acceptable error probabilities, the trial will target 30% as the desirable proportion of patients who are still without progression by radiographic criteria at approximately 6 months (p1=0.30), and will be considered inadequate if only a fraction consistent with 10% are without progression by the same evaluation time (p0=0.10). Initially 12 patients will be enrolled and followed for progression. If 2 or more of the first 12 patients reach 6 months without progression, then enrollment will continue until a total of 35 evaluable patients (37 total patients to allow for a small number of inevaluable patients) have been entered.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have a diagnosis of urothelial carcinoma of the bladder, urethra, ureter, or renal pelvis, with histological confirmation at the Laboratory of Pathology of the NCI (National Cancer Institute), NIH (National Institutes of Health).
* Patients must have progressive metastatic disease. Progressive disease will be defined as new or progressive lesions on cross-sectional imaging. Patients must have at least:
* One measurable site of disease (according to RECIST criteria) that has not been previously irradiated. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation.
* Or, appearance of one new bone lesion.
* Patients must have been previously treated, as defined by the following:
* Treatment with at least one prior cytotoxic agent (which must have included at least one of the following: cisplatin, carboplatin, paclitaxel, docetaxel, or gemcitabine), administered in the perioperative or metastatic setting and may have been administered sequentially (e.g., first-line treatment followed by second-line treatment at time of progression) or as part of a single regimen.
* 18 years of age or older
* ECOG (Eastern Cooperative Oncology Group) performance status of < 2 or Karnofsky Performance Status greater than or equal to 60%
* Resolution of all acute toxic effects of prior chemotherapy, radiotherapy, or surgical procedure to NCI CTCAE (Common Terminology Criteria in Adverse Events) grade less than or equal to 1 or baseline
* Adequate organ function as defined by the following criteria:
* Serum aspartate transaminase (AST (Aspartate transaminase); serum glutamic oxaloacetic transaminase [SGOT (serum glutamic oxaloacetic)]) and serum alanine transaminase (ALT (alanine transaminase); serum glutamic pyruvic transaminase [SGPT (serum glutamic pyruvic transaminase)]) less than or equal to 2.5 times the upper limit of normal (ULN); 5.0 times the ULN in cases of liver metastases
* Total serum bilirubin less than or equal to 1.5 mg/dL (unless elevation from Gilbert's disease or similar syndrome due to slow conjugation of bilirubin)
* Absolute neutrophil count (ANC) greater than or equal to 1000/microL
* Platelets greater than or equal to 100,000/microL
* Serum creatinine less than or equal to 2.0 mg/dl or calculated creatinine clearance (CrCl) greater than or equal to 30 mL/min
* Hemoglobin > 9gm/dL
* PT (prothrombin time), aPTT (activated partial thromboplastin time) must be within normal range
* Patients on anticoagulants may be enrolled as long as the INR (International normalized ratio) does not exceed 3.

EXCLUSION CRITERIA:

* Receipt of an investigational agent within 4 weeks prior to first dose with TRC105
* Major surgery including open biopsy or systemic therapy < 4 weeks prior to first dose with TRC105
* Radiation therapy (except small field) < 3 weeks prior to first dose with TRC105
* Small field radiation therapy < 2 weeks prior to first dose with TRC105
* Minor surgical procedures within 2 weeks
* Uncontrolled chronic hypertension (systolic > 140 or diastolic > 90mm Hg despite optimal therapy)
* Brain metastasis, or leptomeningeal disease because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Unstable angina, MI, symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, DVT (deep vein thrombosis), PTCA (percutaneous transluminal coronary angioplasty) or CABG (coronary artery bypass graft) within the past 6 months
* Cardiac arrhythmias of NCI CTCAE grade greater than or equal to 2 within the last month
* Serious, non-healing wound, ulcer, or bone fracture
* Known active hepatitis
* Hemorrhage within 30 days of dosing or history of persistent gross hematuria
* Known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
* History of hypersensitivity reaction to human or mouse antibody products
* Pregnancy or breastfeeding. Female patients must be surgically sterile (i.e.: hysterectomy) or be postmenopausal, or must agree to use effective contraception during the study and for 3 months following last dose of TRC105. All female patients of reproductive potential must have a negative pregnancy test (serum) within 7 days prior to first dose. Male patients must be surgically sterile or must agree to use effective contraception during the study and for 3 months following last dose of TRC105. The definition of effective contraception will be based on the judgment of the Principal Investigator or a designated associate.
* Other severe acute or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the Investigator would make the patient inappropriate for entry into this study
* History of peptic ulcer disease, unless a subsequent endoscopy has confirmed complete resolution of the ulcer
* History of acquired or inherited hypocoagulopathies (bleeding risk), including but not limited to hereditary hemorrhagic telangiectasis.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B Apolo, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Apolo AB, Karzai FH, Trepel JB, Alarcon S, Lee S, Lee MJ, Tomita Y, Cao L, Yu Y, Merino MJ, Madan RA, Parnes HL, Steinberg SM, Rodriguez BW, Seon BK, Gulley JL, Arlen PM, Dawson NA, Figg WD, Dahut WL. A Phase II Clinical Trial of TRC105 (Anti-Endoglin Antibody) in Adults With Advanced/Metastatic Urothelial Carcinoma. Clin Genitourin Cancer. 2017 Feb;15(1):77-85. doi: 10.1016/j.clgc.2016.05.010. Epub 2016 May 27. PMID 27328856
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0130.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm-TRC105 in Urothelial Carcinoma: TRC 105 every two weeks
  TRC105: 15 mg/kg intravenously
Period: Overall Study
Arm/Group | Single Arm-TRC105 in Urothelial Carcinoma
Started | 13
Completed | 12
Not Completed | 1
Not completed — Refused further treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm-TRC105 in Urothelial Carcinoma
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.28 (6.64)
Gender [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 13
Median Age (Range) [Median (Full Range); unit: years] | 67 [51 to 73]
Karnofsky Performance Status [Number; unit: participants] — Karnofsky Performance Scale: 60 - requires occasional assistance, but is able to care for most of his/her needs; 70 - cares for self, unable to carry on normal activity or to do active work; 80 - normal activity with effort; some signs or symptoms of disease; 90 - able to carry on normal activity; minor signs or symptoms of disease.
  participants
    60 | 1
    70 | 0
    80 | 2
    90 | 10
Primary Tumor Site [Number; unit: participants]
  Bladder | 11
  Upper urinary tract | 2
Metastatic Sites of Disease [Number; unit: participants]
  Lung | 7
  Liver | 2
  Bone | 4
  Any visceral metastases | 10
  Lymph node only | 3
Number of Previous Therapies for Metastatic Disease [Number; unit: participants]
  1 | 3
  2 | 4
  3 | 3
  4 | 2
  5 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Time interval from start of treatment to documented evidence of disease progression. Progressive disease is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (Note: the appearance of one or more new lesions is also considered progression).-
Time Frame: after 6 months on study
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm-TRC105 in Urothelial Carcinoma
Number analyzed (Participants) | 13
Months | 1.9 [1.8 to 2.1]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Single Arm-TRC105 in Urothelial Carcinoma
Number analyzed (Participants) | 13
participants | 12

3. Secondary Outcome: Objective Response
Description: Objective response is defined as the number of participants who meet the criteria for a complete response (CR) or a partial response (PR) per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: up to 25 months
Measure: Number; unit: participants
Arm/Group | Single Arm-TRC105 in Urothelial Carcinoma
Number analyzed (Participants) | 13
participants
  Complete response | 0
  Partial response | 0

4. Secondary Outcome: Median Overall Survival
Description: Date of on-study to the date of death from any cause or last follow up.
Time Frame: up to 25 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm-TRC105 in Urothelial Carcinoma
Number analyzed (Participants) | 13
Months | 8.3 [3.3 to 17.0]

5. Secondary Outcome: Incidence of TRC-105-Related Adverse Events
Description: Adverse events by grade, (e.g. 1 is mild, 2 is moderate, 3 is severe and 4 is life threatening) related to TRC-105.
Time Frame: 24 months
Measure: Number; unit: participants
Groups:
- TRC105 in Urothelial Carcinoma - Adverse Events - All Grades: TRC 105 every two weeks
  TRC105: 15 mg/kg intravenously
  Adverse events grades 1-4 (mild, moderate, severe and life threatening).
- TRC105 in Urothelial Carcinoma - Adverse Events - Grade 1: TRC 105 every two weeks
  TRC105: 15 mg/kg intravenously Grade 1 (mild) adverse events.
- TRC105 in Urothelial Carcinoma - Adverse Events - Grade 2: TRC 105 every two weeks
  TRC105: 15 mg/kg intravenously Grade 2 (moderate) adverse events.
- TRC105 in Urothelial Carcinoma - Adverse Events - Grade 3: TRC 105 every two weeks
  TRC105: 15 mg/kg intravenously Grade 3 (severe) adverse events.
- TRC105 in Urothelial Carcinoma - Adverse Events - Grade 4: TRC 105 every two weeks
  TRC105: 15 mg/kg intravenously Grade 4 (life threatening) adverse events.
Arm/Group | TRC105 in Urothelial Carcinoma - Adverse Events - All Grades | TRC105 in Urothelial Carcinoma - Adverse Events - Grade 1 | TRC105 in Urothelial Carcinoma - Adverse Events - Grade 2 | TRC105 in Urothelial Carcinoma - Adverse Events - Grade 3 | TRC105 in Urothelial Carcinoma - Adverse Events - Grade 4
Number analyzed (Participants) | 13 | 13 | 13 | 13 | 13
participants
  Anemia | 6 | 1 | 4 | 1 | 0
  Anorexia | 1 | 1 | 0 | 0 | 0
  Cough | 1 | 1 | 0 | 0 | 0
  Edema (Limbs) | 1 | 1 | 0 | 0 | 0
  Epistaxis | 6 | 6 | 0 | 0 | 0
  Fatigue | 1 | 1 | 0 | 0 | 0
  Gum bleeding | 4 | 4 | 0 | 0 | 0
  Headache | 9 | 8 | 1 | 0 | 0
  Hematuria | 2 | 1 | 1 | 0 | 0
  Hypoalbuminemia | 1 | 1 | 0 | 0 | 0
  Hypophosphatemia | 2 | 1 | 1 | 0 | 0
  Increased Alanine Aminotransferase | 1 | 1 | 0 | 0 | 0
  Infusion-Related Reaction | 9 | 5 | 4 | 0 | 0
  Maculopapular Rash | 1 | 1 | 0 | 0 | 0
  Nasal Congestion | 3 | 3 | 0 | 0 | 0
  Nausea | 1 | 1 | 0 | 0 | 0
  Proteinuria | 1 | 1 | 0 | 0 | 0
  Skin Infection | 1 | 0 | 0 | 1 | 0
  Telangiectasia | 6 | 6 | 0 | 0 | 0
  Vomiting | 1 | 1 | 0 | 0 | 0
  Xerostomia | 1 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Single Arm-TRC105 in Urothelial Carcinoma
Serious Adverse Events (participants affected / at risk) | 12/13
Other Adverse Events (participants affected / at risk) | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm-TRC105 in Urothelial Carcinoma (N=13)
Bladder infection (Infections and infestations) | 1 (1)
Death NOS (General disorders) | 12 (12)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm-TRC105 in Urothelial Carcinoma (N=13)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 2 (6)
Anemia (Blood and lymphatic system disorders) | 8 (15)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Blurred vision (Eye disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Creatinine increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dental caries (Gastrointestinal disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dizziness (Nervous system disorders) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 5 (11)
Floaters (Eye disorders) | 1 (1)
Flushing (Vascular disorders) | 5 (5)
Gastritis (Gastrointestinal disorders) | 1 (1)
Genital edema (Reproductive system and breast disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (14)
Hematuria (Renal and urinary disorders) | 2 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (6)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Hypotension (Vascular disorders) | 1 (1)
Infusion related reaction (General disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3)
Oral hemorrhage (Gastrointestinal disorders) | 4 (5)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Telangiectasia (Skin and subcutaneous tissue disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No